CLINICAL TRIAL: NCT01870622
Title: Confirmation of Correct Tracheal Tube Placement in Newborn Infants - a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00036974
Record Dates: First submitted 2013-05-29; First posted 2013-06-06 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Newborn Infant
Keywords: Newborn,; Infant,; Endotracheal Intubation,; Carbon dioxide detector,; Flow waves

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ECO2 (Active Comparator): ECO2 will be used to confirm correct tube placement in newborn infants.
  Interventions: Procedure: ECO2
- Flow waves (Experimental): Flow waves will be used to confirm correct tube placement
  Interventions: Procedure: Flow waves

INTERVENTIONS:
Procedure: Flow waves — Flow waves will be used to confirm correct tube placement in newborn infants.
  Arms: Flow waves
Procedure: ECO2 — ECO2 will be used to confirm correct tube placement in newborn infants.
  Arms: ECO2

SUMMARY:
Most premature babies have difficulty breathing at birth and need help (resuscitation). The treatment for this is to gently inflate their lungs with a resuscitation device and a facemask. To gently inflate an infant's lungs the clinical team places a breathing tube in the windpipe and blow air into your baby's lung (puffs). With the first puffs the clinical team checks if the breathing tube is correctly placed within the windpipe. The investigators routinely use a detector which checks for exhaled carbon dioxide or the graphical display of waves forms of the infants breathing to check that the breathing tube position. However, the investigators do not know which one (exhaled carbon dioxide or the graphical display of waves forms) is better to check that the breathing tube position is correct and therefore the investigators would like to study them. The purpose of this study is to compare exhaled carbon dioxide detectors (ECO2 group) with the graphical display of waves forms (flow waves group) to provide us with information on how the investigators can help babies who struggle with breathing at birth.

ELIGIBILITY:
Inclusion Criteria:

* All infants (term and preterm) born at The Royal Alexandra Hospital who require endotracheal intubation in the delivery room or neonatal intensive care unit will be recorded.

Exclusion Criteria:

* Infants will also be excluded if their parents refuse to give consent to this study.

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Using flow waves will increase the percentage of correct tube placement in newborn infants | within the first 10 inflations
  Flow waves and exhaled Carbon dioxide will be compared using the numbers of inflation needed to identify correct tube placement.
  We will compare the number of inflation in each group to identify which device can identify correct tube placement faster and more accurately.
  Outcome will be number of inflation until correct tube placement has been identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Schmolzer GM, O'Reilly M, Davis PG, Cheung PY, Roehr CC. Confirmation of correct tracheal tube placement in newborn infants. Resuscitation. 2013 Jun;84(6):731-7. doi: 10.1016/j.resuscitation.2012.11.028. Epub 2012 Dec 1. PMID 23211476
- [Background] Schmolzer GM, Poulton DA, Dawson JA, Kamlin CO, Morley CJ, Davis PG. Assessment of flow waves and colorimetric CO2 detector for endotracheal tube placement during neonatal resuscitation. Resuscitation. 2011 Mar;82(3):307-12. doi: 10.1016/j.resuscitation.2010.11.008. Epub 2010 Dec 16. PMID 21167628
- [Background] Schmolzer GM, Hooper SB, Crossley KJ, Allison BJ, Morley CJ, Davis PG. Assessment of gas flow waves for endotracheal tube placement in an ovine model of neonatal resuscitation. Resuscitation. 2010 Jun;81(6):737-41. doi: 10.1016/j.resuscitation.2010.02.018. Epub 2010 Mar 23. PMID 20334964
- [Background] Aziz HF, Martin JB, Moore JJ. The pediatric disposable end-tidal carbon dioxide detector role in endotracheal intubation in newborns. J Perinatol. 1999 Mar;19(2):110-3. doi: 10.1038/sj.jp.7200136. PMID 10642970
- [Background] Hosono S, Inami I, Fujita H, Minato M, Takahashi S, Mugishima H. A role of end-tidal CO(2) monitoring for assessment of tracheal intubations in very low birth weight infants during neonatal resuscitation at birth. J Perinat Med. 2009;37(1):79-84. doi: 10.1515/JPM.2009.017. PMID 18976048
- [Background] O'Donnell CP, Kamlin CO, Davis PG, Morley CJ. Endotracheal intubation attempts during neonatal resuscitation: success rates, duration, and adverse effects. Pediatrics. 2006 Jan;117(1):e16-21. doi: 10.1542/peds.2005-0901. PMID 16396845
- [Background] Leone TA, Rich W, Finer NN. Neonatal intubation: success of pediatric trainees. J Pediatr. 2005 May;146(5):638-41. doi: 10.1016/j.jpeds.2005.01.029. PMID 15870667